CLINICAL TRIAL: NCT05441540
Title: Internal Jugular Vein Compression Collar for Novel Symptomatic Treatment of Venous Pulsatile Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-3127
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2023-02

CONDITIONS: Pulsatile Tinnitus
Keywords: pulsatile tinnitus; Internal Jugular Vein (IJV) collar
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: All participants will be in a single treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Device will be fitted and worn up to two hours daily and participants will log changes in symptom intensity before and during device usage
  Interventions: Device: Internal Jugular Vein Compression Collar

INTERVENTIONS:
Device: Internal Jugular Vein Compression Collar — The current FDA approved internal jugular vein compression collar, marketed as the Q collar, is manufactured by Q30 Innovations Home. It is designed to be worn around the neck of individuals aged 13 and older. It functions by lightly compressing the internal jugular vein's bilaterally, safely increasing intracranial volume and intracranial pressure. The FDA approved neck collar device is made of a thermoplastic elastomer that is specifically fitted to an individual to provide mild internal jugular vein compression. The product was developed and confirmed with ultrasonography to confirm appropriate fit and compression of the vein based on an athlete's neck circumference.
  Other Names: Q collar

SUMMARY:
This study seeks to pilot an evaluation of whether an external jugular vein compression collar approved by the US Food and Drug Administration (FDA) for contact sports can provide symptomatic relief of venous pulsatile tinnitus. Furthermore, the study will evaluate quality of life impacts of the device and adherence by users.

DETAILED DESCRIPTION:
Background: Tinnitus is a medical condition with a wide variety of causes that is characterized by the perception of sound, often described as ringing or buzzing, without an external stimulus. Venous pulsatile tinnitus is a specific subtype of tinnitus with limited treatment options: some cases can be treated with surgical correction of an underlying vascular defect, others are entirely idiopathic. The clinical diagnostic hallmark of venous pulsatile tinnitus is relief of symptoms with light compression of the ipsilateral external jugular vein by the physician. Internal jugular vein compression collars, FDA approved devices currently used to prevent brain injuries in contact sports, function by this exact same method. Therefore, it is believed that these collars can treat pulsatile tinnitus.

Study Design:

This is a non-blinded, interventional, prospective single cohort pilot study that will recruit 20 patients diagnosed with pulsatile tinnitus at the UNC Meadowmont Ear Nose and Throat (ENT) clinic (see methods for inclusion/exclusion criteria). Volunteers will compare tinnitus intensity before and after administration of the collar, take the collar home and evaluate its symptomatic efficacy over a 2-4-week period, and return to clinic to complete data on quality of life and longitudinal impacts. This data will be analyzed for significance.

Expected Outcomes:

It is expected that collar administration will offer immediate symptomatic relief, illustrated as significant improvement on the tinnitus intensity scale during their initial clinic visit Symptomatic improvement will be sustained while wearing the collar, measured by sustained improvement in the tinnitus handicap inventory over the course of the study. Lastly, the collar will improve quality of life as measured by patient reported outcome scales administered pre and post participation.

ELIGIBILITY:
Inclusion Criteria

* Male or female age 18 years and older
* Diagnosis of venous pulsatile tinnitus
* Patient at UNC ENT Meadowmont Clinic

Exclusion Criteria

* Increased presence of acid in the body or excessive blood alkalinity
* Open head injury (including in or around the eye) within the past six months
* Pseudotumor cerebri (false brain tumor)
* Presence of brain or spinal shunt
* Known seizure disorder
* Known airway obstruction
* Increased likelihood of blood clotting (coagulation)
* Skin injury, rash, or other abnormality on or around the neck
* age <18
* unable to provide written consent,
* history of neurological deficits,
* previous cerebral infarction (blockage or narrowing in the arteries supplying blood and oxygen to the brain)
* severe head trauma
* medical contraindications to restriction of blood outflow via the internal jugular veins
* glaucoma (narrow angle or normal tension - increased pressure in the eyes),
* hydrocephalus (increased fluid on the brain)
* recent penetrating brain trauma (within 6 months),
* known carotid hypersensitivity
* known increased intracranial pressure
* idiopathic intracranial hypertension
* known intracranial vascular malformation (e.g. aneurysm, arteriovenous malformation, cavernoma)
* central vein thrombosis
* not tolerating initial fitting of collar.
* Known pregnancy (this is not a direct contraindication but is being made out of an abundance of caution)
* Inability to speak or comprehend English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S Succop, B.S., Principal Investigator — Medical Student; Brian Sindelar, MD, Study Director — brian_sindelar@med.unc.edu
Locations (1):
- UNC Meadowmont ENT Clinic, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 to 36 months following publication
Access Criteria: see above

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 20
Completed | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 15
  Race/Ethnicity: Black/African American | 2
  Race/Ethnicity: Other Race | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Height and weight were obtained using the most recent data available from the medical record.
  The BMI categories are: Underweight = <18.5; Normal weight = 18.5-24.9; Overweight = 25-29.9; Obesity = BMI of 30 or greater.
  kg/m^2 | 26 (3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pulsatile Tinnitus Symptom Intensity
Description: Assessing the difference in pulsatile tinnitus symptom intensity without the collar vs. with the collar as evaluated by a 10 point Likert scale ranging 0-10 where 0 is no symptoms and 10 is maximal symptom intensity. Participants were allowed to use the collar for up to 30 days as often or as little as desired on a weekly basis but no longer than 2 hours continuously in accordance with the collar's FDA clearance. Participants completed a survey for each day of use reporting the intensity of their symptoms before wearing the collar and while wearing the collar. The difference between these symptom intensities with and without the collar is a single data point. Each data point was aggregated across all participants and across all days of use. From these aggregated data, the median and interquartile range were calculated. Therefore, the outcome is the median difference in intensity before and during wear of every day of collar use by every participant.
Time Frame: From immediately before collar placement to less than or equal to two hours of wearing the collar for each day of use.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 18
units on a scale | 3 [1 to 4]
Statistical Analysis 1: Comparison: Treatment Group; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline in Tinnitus Quality of Life From Collar Usage
Description: Determine if quality of life changes appreciably while using the collar and participating in the study as measured by the tinnitus handicap inventory (THI), a 25-item validated survey that evaluates the degree of impact a patient's tinnitus has on their quality of life. It is scored on a scale of 0-100, where 0 represents no handicap and 100 represent catastrophic handicap.
Time Frame: Baseline, 5 weeks later upon completion of study participation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 18
score on a scale | 12 [7 to 16]
Statistical Analysis 1: Comparison: Treatment Group; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Temporality of Collar Usage Effect on Symptom Intensity
Description: Participants were allowed to use the collar for up to 30 days as often or as little as desired on a weekly basis but no longer than 2 hours continuously in accordance with the collar's FDA clearance. Participants completed a survey containing a 0-10 point Likert scale of tinnitus intensity (where 0 is no symptoms and 10 is maximal symptom intensity) for each day of use reporting the intensity of their symptoms before wearing the collar and while wearing the collar. The difference between these symptom intensities with and without the collar is a single data point. These data points were grouped by week (week 1, week 2, week 3, week 4) across participants and the median for each reported. These medians were compared statistically to determine if the effect of the collar on symptom intensity changed by week.
Time Frame: From immediately before collar placement to less than or equal to two hours of wearing the collar for each day of use.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 18
units on a scale
  Week 1 | 2 [1.00 to 3.00]
  Week 2 | 2 [2.00 to 3.00]
  Week 3 | 2 [1.00 to 3.00]
  Week 4 | 3 [1.25 to 3.00]
Statistical Analysis 1: Comparison: Treatment Group; Test type: Other; p = 0.7613, Kruskal-Wallis

4. Secondary Outcome: Observed Clinical Effect of Collar vs. Home Use Effect of Collar
Description: Assessing the difference in pulsatile tinnitus symptom intensity without the collar vs. with the collar as evaluated by a 10 point Likert scale ranging 0-10 where 0 is no symptoms and 10 is maximal symptom intensity. Participants were allowed to use the collar for up to 30 days as often or as little as desired on a weekly basis but no longer than 2 hours continuously in accordance with the collar's FDA clearance. Participants completed a survey for each day of use reporting the intensity of their symptoms before wearing the collar and while wearing the collar. The difference between these symptom intensities with and without the collar is a single data point. Each of these data points were grouped by location of measurement (in clinic vs. at-home) across participants, the medians of each of these two groups were reported, and then statistically compared to evaluate if the change in symptom intensity varied by location of measurement.
Time Frame: From immediately before collar placement to less than or equal to two hours of wearing the collar for each day of use.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 18
units on a scale
  Clinic Measurement | 2 [1.00 to 3.00]
  Home Measurement | 3 [2.00 to 3.00]
Statistical Analysis 1: Comparison: Treatment Group; Test type: Other; p = 0.7640, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through the study debrief visit, a total of about 5 weeks.
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT05441540/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT05441540/ICF_000.pdf